CLINICAL TRIAL: NCT01391052
Title: Pretreatment With Norethindrone Acetate Prior to Levonorgestrel IUS Insertion for Heavy Menstrual Bleeding
Acronym: Mirena IUD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scott and White Hospital & Clinic (Other)
Responsible Party: Patricia Sulak, MD/principal investigator, Scott and White Hospital & Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90378
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-01

CONDITIONS: Heavy Menstrual Bleeding; Menorrhagia; Hypermenorrhea
Keywords: Intrauterine system; reproductive age; menstrual bleeding
MeSH Terms: conditions — Menorrhagia | interventions — Norethindrone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Norethindrone acetate pretreatment (Active Comparator): This arm will receive two cycles of norethindrone acetate before LVN IUS insertion.
  Interventions: Drug: Norethindrone acetate pretreatment
- No pretreatment (Other): LVN IUS is placed without norethindrone acetate pretreatment.
  Interventions: Other: No pretreatment

INTERVENTIONS:
Drug: Norethindrone acetate pretreatment — 5 mg tablets, three times a day for 21 days for 2 menstrual cycles.
  Other Names: Aygestin
  Arms: Norethindrone acetate pretreatment
Other: No pretreatment — LVN IUS is placed withour Norethindrone acetate pretreatment.
  Arms: No pretreatment

SUMMARY:
Problematic uterine bleeding after the insertion of the LNG IUS is a well documented side effect. The levonorgestrel intrauterine system (LNG IUS) was approved for treatment of heavy menstrual bleeding (HMB) by the FDA in October 2009. To reduce the incidence and severity of post-insertional uterine bleeding, pretreatment with norethindrone acetate may effectively slough the endometrium prior to insertion of the LNG IUS.

DETAILED DESCRIPTION:
This study will examine whether or not pretreatment with oral norethindrone acetate prior to the insertion of a hormonal intrauterine device will affect post-insertional uterine bleeding. The subjects enrolling in the study will have documented heavy menstrual bleeding (HMB) and desire the levonorgestrel intrauterine system (LNG IUS) (Mirena®, Bayer, Inc. Pittsburgh, PA) for symptomatic relief. HMB for this study is defined as heavy bleeding at regular intervals at least 20-40 days apart. Subjects will be randomized to one of two groups. One group will receive norethindrone acetate for two consecutive months prior to LNG IUS insertion while the other group will proceed with direct insertion of the LNG IUS with no hormonal pre-treatment. Subjects will be followed for a period of 180 days post LNG IUS insertion. Bleeding patterns will be recorded daily.

ELIGIBILITY:
Inclusion Criteria:

* You must be between 18-45 years old
* You have Heavy Periods

Exclusion Criteria:

* You are pregnant
* You are currently using hormonal contraception or hormonal therapy
* You have a history of pelvic inflammatory disease (and have not had a normal pregnancy since)
* You had an infected abortion within the last three months
* You have abnormal or cancerous cells of the cervix or uterus
* You have an actine infection in your genital organs
* Known or suspected breast cancer
* Active liver disease or tumors
* Allergy to levonorgestrel or norethindrone
* You currently have deep vein thrombosis, pulmonary embolism, or history of these conditions
* you currently have active or recent (within the past year) arterial thromboembolic disease (such as a stroke or myocardial infarction) these conditions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Total number of bleeding days | up to 180 days
  Number of days on study calendars with menstrual flow

SECONDARY OUTCOMES:
Menorrhagia Questionnaire | up to 180 days
  Patients will assess the impact of their menstrual bleeding on their lifestyle.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J Sulak, MD, Principal Investigator — Scott and White Hospital & Clinic
Locations (1):
- Scott and White Hospital and Clinic, Temple, Texas, United States